CLINICAL TRIAL: NCT06928948
Title: Medium-term Results of the LPS™ System for Segmental Resection of the Distal Femur, a Multicenter Retrospective Study.
Brief Title: Medium-term Results of the LPS™ System for Segmental Resection of the Distal Femur, a Multicenter Retrospective Study (RESIF)
Acronym: RESIF
Status: Enrolling by invitation | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC24.0294 - RESIF
Record Dates: First submitted 2025-02-13; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2024-10

CONDITIONS: Prosthesis Failure
Keywords: megaprosthesis; knee replacement
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Femur replacement — Reconstruction using the Limb Preservation System™ for segmental resection of the distal femur.

SUMMARY:
The reconstruction of the distal femur using modular systems has become increasingly popular over the years, surpassing primary arthrodesis or amputation. Despite the significant advantages of using megaprostheses, complications are not uncommon. Although the Limb Preservation System™ (LPS™, DePuy Synthes; Warsaw, USA) is one of the most widely used megaprostheses in the French market, there is currently no national evaluation of this system, and only two studies have been conducted worldwide.

The aim of our study is to present the mid-term survival rates of the LPS™ implant in order to answer three main questions:

1. What are the overall outcomes of the LPS™ system in distal femur replacement?
2. What factors are associated with a reduced survival rate of the implant?
3. What is the cumulative risk of complications according to Henderson's classification?

The secondary objective is to analyze the occurrence of specific failures, providing insights for potential improvements in the design and use of the LPS™ implant.

ELIGIBILITY:
Inclusion Criteria:

- Patients who underwent distal femoral reconstruction using the LPS system.

Exclusion Criteria:

* Lost to follow-up before 3 months.
* Associated tibial reconstruction using the LPS system.
* Total femoral reconstruction using the LPS system.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The institutional databases of university hospitals belonging to the HugOrtho network (Hôpitaux Universitaires du Grand Ouest) will be examined to identify patients who will have undergone reconstruction using the Limb Preservation System™ (LPS™, DePuy Synthes; Warsaw, USA) for segmental resection of the distal femur, regardless of the indication.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
LPS stent failure | From enrollment to last consultation
  Failure will be defined as the replacement of the femoral anchorage or amputation.

SECONDARY OUTCOMES:
complications of the LPS stent | From enrollment to last consultation
  Complications will be defined according to Henderson's classification.
Surgical revision of the LPS stent | From enrollment to last consultation
  Any reoperation on the knee after the LPS one

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement